CLINICAL TRIAL: NCT03612999
Title: Data Acquisition to Model Glycemic Response to Food and Other Events Using Real-Time Continuous Glucose Monitoring (RT-CGM)
Brief Title: Data Acquisition to Model Glycemic Response
Acronym: SDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Savvysherpa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Pro00022817
Record Dates: First submitted 2018-07-23; First posted 2018-08-02 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2020-09

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- CGM and Activity Tracker (Experimental): Subjects receive a continuous glucose monitor (CGM) and activity tracker and are instructed to record daily activities and psychological data.
  Interventions: Device: Dexcom continuous glucose monitor; Device: Fitbit activity tracker; Behavioral: Subjects record daily activity; Behavioral: Subjects record psychological state

INTERVENTIONS:
Device: Dexcom continuous glucose monitor — Continuous glucose monitors (CGMs) record subjects glucose levels
Device: Fitbit activity tracker — Activity trackers will record subjects' physical activity, heart rate, and sleep.
Behavioral: Subjects record daily activity — Subjects will record their daily activities, either on paper or on a secure texting app.
Behavioral: Subjects record psychological state — Subjects will record their psychological state, either on paper or on a secure texting app.

SUMMARY:
To learn about individual glycemic response to physiological and psychological conditions across a diverse population, the investigators will collect sensor and lifestyle data directly from participants as they engage in daily activities. The investigators will collect real-time glucose data from a continuous glucose monitor (CGM) system; accelerometer, aggregated activity, and sleep data from a wrist-worn activity tracker; mood and experiential data; and food information. Non-sensor data will be collected using a paper log, or via a study app when available.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years old
* Be able to read, speak, and understand English
* Have a primary care provider

Exclusion Criteria:

* Not receive or require kidney dialysis
* Not be pregnant
* Not have type 1 diabetes
* Not have type 2 diabetes and be prescribed three or more daily injections of insulin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2020-09-23 (Actual); Study Completion 2020-09-23 (Actual)

PRIMARY OUTCOMES:
Glucose Level (mg./dl.) | 20 days per participant
  Estimated glucose concentration (mg./dl.) sampled every five minutes by a continuous glucose monitor (CGM).

SECONDARY OUTCOMES:
Activity level (steps per hour) | 20 days per participant
  Activity level (steps per hour) as determined from data from wrist-worn accelerometer
Food Consumption (type and quantity) | 20 days per participant
  Food items as described by user in food logs, along with time of consumption.
Activities of daily living (free form) | 20 days per participant
  Participants may log any activity of daily living they choose, including social interactions, house work, and leisure activities. Activities are described by users and logged in interval form with start-time and end-times.
Psychological state (free-form) | 20 days per participant
  Participants may log any psychological information they choose including mood, energy level, or cognitive function. Psychological states are described by users and logged with time or interval in which that psychological state was experienced.
Sensor wear time (wear / no-wear intervals) | 20 days per participant
  Participants will log intervals in which they are and are not wearing the CGM over the course of their participation in the study.
Transmitter life expectancy (number of minutes) | 20 days per participant
  In cases where participants wear sensors until the end of the transmitter's life, the number of minutes transmitter was operational.

CONTACTS AND LOCATIONS:
Locations (1):
- Savvysherpa, LLC, Minnetonka, Minnesota, United States